CLINICAL TRIAL: NCT02143011
Title: Synergistic Effects of Stress and Sugar Feeding on Metabolism
Brief Title: Stress and Sugar Synergy
Acronym: SSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of California, San Francisco (Other); USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 574149
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Metabolic Syndrome; Insulin Resistance; Dyslipidemia
Keywords: sugar; sucrose; fruit juice; orange juice; metabolism; immune cell aging; lipids
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Dyslipidemias | interventions — Sucrose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- orange juice (Other): no sugar
  Interventions: Other: orange juice; Other: sucrose
- sugar beverage (Other): no sugar
  Interventions: Other: orange juice; Other: sucrose

INTERVENTIONS:
Other: orange juice — intervention assigned: 2-week consumption of naturally-sweetened orange juice providing 25% of energy requirement
Other: sucrose — intervention assigned: 2-week consumption of sucrose-sweetened beverage providing 25% of energy requirement

SUMMARY:
The main objectives of this study are to test the hypotheses that: 1) consumption of beverages sweetened with sucrose will increase risk factors for cardiovascular disease to a greater extent than a naturally-sweetened fruit juice such as orange juice, and 2) chronic psychological stress may augment the adverse metabolic effects of sugar intake. The study intervention consists of 2-week's consumption of 25% of energy as sugar provided either as a sucrose-sweetened beverage or naturally-sweetened orange juice.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 28-35
* Self report of stable body weight during the past six months
* High stress participants: Perceived Stress Scores (PSS) ≥ 24, and the presence of a predefined chronically stressful event as assessed by the Telephone screening questions. (IDS scores are not an inclusion criteria in this group, merely a rule-out for the low stress participants).
* Low stress participants: PSS scores ≤ 8, Inventory for Depressive Symptom (IDS) scores ≤ 14, and the absence of any predefined chronically stressful events as assessed by the telephone screening questions.

Exclusion Criteria:

* glucose intolerance
* Evidence of liver disorder
* Evidence of kidney disorder
* Evidence of thyroid disorder
* Systolic blood pressure consistently over 140mmHg or diastolic blood pressure over 90mmHg
* Triglycerides > 200mg/dl
* LDL-C > 130mg/dl
* Hemoglobin < 8.5 g/dl
* pregnant or lactating women
* Current, prior (within 12 months), or anticipated use of any hypolipidemic or anti-diabetic agents
* Use of Selective Serotonin Reuptake Inhibitors and anti-hypertensive medications
* Any other condition that, in the opinion of the investigators, would put subject at risk
* Strenuous exerciser
* surgery for weight loss
* Diet exclusions: food allergies, special dietary restrictions, habitual ingest of >2 alcoholic beverages/day

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
24-hour triglyceride area under the curve | Baseline and 2-week intervention
  28 serial blood samples are collected over a 24 hour period.

SECONDARY OUTCOMES:
Markers of immune cell aging | Baseline and 2-week intervention

OTHER OUTCOMES:
3 hour oral glucose tolerance test | Baseline and 2-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Peter Havel, D.V.M, Principal Investigator — University of California, Davis; Kimber Stanhope, Ph.D, R.D., Study Director — University of California, Davis
Locations (1):
- Clinical Research Center, Sacramento, California, United States